CLINICAL TRIAL: NCT02344082
Title: Pharmacists Provide Telemedicine in Addition to Clinic Visits to Improve Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00051947; 1819 (Other: Other)
Record Dates: First submitted 2015-01-08; First posted 2015-01-22 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Telemedicine
MeSH Terms: interventions — Telemedicine

ARMS (2):
- Standard of Care (No Intervention): The control arm will receive face-to-face pharmacy clinic visits per usual care.
- Intervention Arm (Active Comparator): The intervention arm will receive pharmacy clinic visits plus additional telephone follow-up.
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — The intervention arm will receive pharmacy clinic visits plus additional telephone follow-up.
  Arms: Intervention Arm

SUMMARY:
This prospective study will include both an intervention and control arm. The control arm will receive face-to-face pharmacy clinic visits per standard of care. The intervention arm will receive pharmacy clinic visits plus additional telephone follow-up. Patients with a hemoglobin A1c in the last 3 months greater than 9% will be eligible. Eligible patients must have a primary care physician at Johns Hopkins Outpatient Center (JHOC) or East Baltimore Medical Center (EBMC).

Purpose: To compare the change in hemoglobin A1c over the 3 month study period in the intervention group in which patients participate in telemedicine, to a control group in which they do not

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a primary care provider at JHOC or EMBC
* Patients have seen primary care provider within last 6 months
* Patients with hemoglobin A1c greater than 9%

Exclusion Criteria:

* Patients <18 years of age
* Patients with previously established care with JHH ambulatory care pharmacist
* Patients with communication barriers who do not have a caregiver
* Patients with new diagnosis of diabetes
* Patients who are pregnant or planning to become pregnant during the time of the study
* Patients followed by Endocrinology or Diabetes Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c | 3 months
  A1c at 3 months - A1c at Baseline

SECONDARY OUTCOMES:
Patient adherence to office visits (# visits attended/# of visits scheduled) | 3 months
  # visits attended/# of visits scheduled
Pharmacist interventions (Number of pharmacist interventions (lifestyle or medication changes) made) | 3 months
  Number of pharmacist interventions (lifestyle or medication changes) made
Patient satisfaction (Based on survey results) | 3 months
  Based on survey results at final pharmacy clinic visit
Telemedicine in Usual Care (Percent of patients who receive telephone call under usual care) | 3 months
  Percent of patients who receive telephone call under usual care
Telemedicine Adherence (Percent of telephone encounters completed in intervention arm) | 3 months
  Percent of telephone encounters completed in intervention arm